CLINICAL TRIAL: NCT05706779
Title: Combination of Encorafenib Plus Cetuximab in a Neoadjuvant Setting in Patients With Braf v600e-mutates Localised Colon or Upper Rectum Cancer (Neoraf Study)
Brief Title: Encorafenib Plus Cetuximab in a Neoadjuvant Setting in Patients With BRAF Mutation Localised Colon or Upper Rectum Cancer
Acronym: NEORAF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: Pierre Fabre Laboratories (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFCD 2006 NEORAF
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer; BRAF V600E Mutation Positive
MeSH Terms: conditions — Colorectal Neoplasms | interventions — encorafenib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Encorafenib + Cetuximab (Experimental)
  Interventions: Drug: Encorafenib Oral Capsule + Cetuximab

INTERVENTIONS:
Drug: Encorafenib Oral Capsule + Cetuximab — Encorafenib: 4 capsules 75 mg/day (300 mg) , 7 days/7 during 6 weeks Cetuximab: 500mg/m2 intravenous route every 2 weeks (D1, D14, D28), for 3 cycles over 4 weeks.

SUMMARY:
This is a pilot trial which aims to assess the concept of anti-BRAF neoadjuvant treatment (encorafenib) in combination with cetuximab in patients with colon cancer or rT3/T4 supra-peritoneal upper rectal cancer based on a pre-operative CT-scan. About 10% of patients will have a mutated BRAF V600E tumour and the objective is to include 30 patients with this mutation.

If the tumour is not confirmed as a carrier of the BRAF V600E mutation or has an RAS mutation according to centralised assessment, treatment will be discontinued in this patient and cancer surgery will be organised as soon as possible. The patient will be excluded from the statistical analysis and will be replaced by a new patient in order to obtain 30 patients with confirmed BRAF V600E mutation and RAS wild type . It should be noted that less than a 3% discrepancy between the numbers of local laboratory results and central analysis results, has been reported in over 600 BRAF V600E mutated colon cancers in the BEACON CRC study. Based on these figures, there should be 0 or 1 patient with discrepant results in the study presented here.

Furthermore, in the hypothetical case of a patient who is an early permanent discontinuation of the study prior to surgery, this patient will be replaced in order to obtain a total of 30 patients who underwent surgery after neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed and dated by the patient and the investigator
* Age ≥18 years at time of informed consent
* Adenocarcinoma of the colon or of the upper rectum (supra-peritoneal) considered operable and histologically confirmed, localised, mutated BRAF V600E determined in a biopsy specimen and resectable after CT-scan assessment.

Remark: Centralised analysis of BRAF status will be performed in order to confirm the existence of the mutation concomitantly with the 1st cycle of therapy

* Tumour stage rT4 or rT3 with ≥ 5 mm extra-mural extension in a CT-scan.

  * rT3 with high risk: Tumour spread from the peripheral serosa and extension to the adjacent peritoneal fat of more than 5 mm in its longest diameter (both axial and coronal planes)
  * rT4: Extension to an adjacent organ
* Patient able to provide a sufficient quantity of representative tumour sample (slides or extracted tumor DNA) for centralised analysis of RAS and BRAF mutational status.
* WHO performance status 0 or 1
* Haematological function considered satisfactory:

  * Polymorphonuclear neutrophils (PMN) ≥ 1,500/mm3
  * Platelets ≥ 100,000/mm3
  * Hb ≥ 9g/dL
* Creatinine clearance > 50 mL/min (according to MDRD formula).
* Serum levels of magnesium within normal limits of the centre.
* Total serum bilirubin ≤ 25 μmol/L, ALT and/or AST ≤ 2.5 x ULN.
* Cardiac function considered satisfactory:

  o Corrected mean QT interval for heart rate according to the Fridericia formula (QTcF) ≤ 480 ms.
* Patient able to take medicinal products by mouth (OD).
* Female Patients postmenopausal for at least one year or surgically infertile for at least 6 weeks, or effective contraception for male and female patients of childbearing potential for 2 months after the end of the investigational treatments
* A negative pregnancy test for inclusion for all female patients of child-bearing FFCD 2006 - NEORAF Version 1.0- 21/October2022 Page 7 of 69 potential.
* Patient covered by a plan of the French Social Security system

Exclusion Criteria:

* Existence of distant metastases or adjacent nodules of peritoneal carcinosis (M1).
* Existence of a dual-tumour location.
* known RAS mutation
* Peritonitis (secondary to perforation of the tumour) or symptomatic colonic occlusion or a temporary colostomy to prevent a sub-occlusion.
* Patient in whom an indication for radiotherapy exists based on the multidisciplinary meeting/board pre-operatively.
* Previous treatment with a BRAF inhibitor, cetuximab or other anti-EGFR treatment.
* History of acute or chronic pancreatitis within the 6 months prior to start of the study treatment.
* A history of chronic inflammatory bowel disease requiring treatment (with immuno-modulators or immuno-suppressants) ≤ 12 months before start of study treatment.
* Patient with decreased cardiovascular function or clinically significant cardiovascular disease:

  1. History of myocardial infarction, acute coronary syndrome (including unstable angina, coronary artery bypass grafting, coronary angioplasty or stent placement) ≤ 6 months prior to start of the study treatment.
  2. Symptomatic congestive heart failure (CHF) (grade 2 or higher), history or current evidence of cardiac arrhythmia and/or a clinically significant conduction disorder ≤ 6 months prior to start of the study treatment, except atrial fibrillation with controlled heart rate and paroxysmal supra-ventricular tachycardia.
* Child-Pugh class B or C cirrhosis.
* Deterioration of gastro-intestinal function or a disease which may significantly impair the absorption of encorafenib, e.g.: ulcer disease, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome, small bowel resection
* A previous or concomitant malignant tumour within 5 years prior to the study. Except for basal cell or squamous skin cancer, superficial cancer of the bladder, intra-epithelial carcinoma of the prostate, carcinoma in situ of the uterine cervix or any other malignant tumour which has been treated adequately and which has not recurred during the three years prior to entry in the study.
* A concomitant neuro-muscular disease associated with high levels of creatinine kinase (CK).

Remark: inflammatory muscular disease, muscular dystrophy, amyotrophic lateral sclerosis (ALS), spinal muscular atrophy.

* History of infection with human immunodeficiency virus (HIV).
* Active infection with hepatitis B or hepatitis C.
* Known existence of Gilbert syndrome
* Use of medicinal plants/dietary supplements or other medicinal products or foods that are potent inducing agents or inhibitors of cytochrome P450 (CYP) 3A4/5 ≤ 1 week before start of the study treatment.
* Known severe hypersensitivity reactions to monoclonal antibodies or BRAF-inhibitors (grade ≥ 3), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
* Participation in a clinical study with administration of an investigational product within 4 weeks or five times the half-life of the investigational product, according to the longest period, prior to the first dose of the study treatment.
* Persons who are deprived of their freedom or who are under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
To assess the rate of significant tumour regression (TRG 0 to 2 according to Ryan's modified score of the AJCC 2010) | 6 months after completing inclusions
  with centralised review after neoadjuvant treatment with encorafenib and cetuximab, in patients with RAS wild type localised colon or upper rectum cancer (CC) and carriers of the BRAF V600E mutation.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Gallois, MD, Principal Investigator — Paris HEGP
Locations (1):
- Chu - Hôpital Européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: No